CLINICAL TRIAL: NCT06790069
Title: Safety and Feasibility of the Integration of Ada Into the Mobile MomConnect Information Service for Pregnant Women and New Mothers in South Africa
Brief Title: Evaluating the Impact of a Symptom Checker on Healthcare-seeking Decisions: a Mixed-Methods Study
Acronym: SAFEMOM
Status: Completed | Type: Observational
Sponsor: Ada Health GmbH (Industry)
Collaborators: Reach Digital Health (formerly Praekelt.org) (Unknown); Citizen Surveys (Unknown); Rockefeller Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: StAP0012
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Maternal Health Care
Keywords: maternal health; mobile health tools; symptom checker

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to evaluate the integration of a symptom checker (SC) into the MomConnect (MC) platform to support maternal healthcare in South Africa. The main questions it aims to answer are:

* Does the SC provide safe and appropriate medical advice?
* Does the SC help mothers make informed decisions about when and where to seek healthcare, saving time and money by avoiding unnecessary visits?
* Does the SC improve access to care for those facing significant healthcare barriers?

Participants will answer survey questions before and after using the SC. A subset of participants will also be invited to participate in structured telephone interviews.

The study will help researchers assess the SC's impact on healthcare decisions and resource use in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Women registered with MomConnect, who would like to assess their or their child's symptoms
* At least 18 years of age
* Women with access to WhatsApp
* Capable of completing a symptom assessment in English

Exclusion Criteria:

* Incapable of completing a symptom assessment in English via WhatsApp (e.g. due to illiteracy, language barrier, mental impairment or inebriation or other incapacity or lack of access to WhatsApp)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of users of MomConnect a program developed by the National Department of Health (NDOH) in South Africa and Reach Digital Health for pregnant women and young mothers.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Proportion of appropriate advice by the SC for mother and child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.
Proportion of safe advice by the SC for mother and child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.

SECONDARY OUTCOMES:
Potential prevention of a health problem in Perinatal Period for Mother or Child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.
Potential prevention of a SEVERE health problem in Perinatal Period for Mother or Child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.
Potential Occurrence of a health problem (adverse event) in Perinatal Period for Mother and Child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.
Potential Occurrence of a SEVERE health problem (severe adverse event) in Perinatal Period for Mother or Child | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment.
Health seeking behaviour before and after using Ada+MomConnect | From data collection with participant enrolment to the completion of the follow-up survey send out 1 week after enrolment.
Number of participants who consulted an HCP after using Ada+MomConnect | After completion of the follow-up survey send out 1 week after enrolment.
Gaining of health information in a fast and standardised way | On the day of enrolment.
Usability | On the day of enrolment.
Time saved from avoiding unnecessary healthcare consultations | On the day of enrolment.
Time saved and associated estimate of income retained through avoiding unnecessary healthcare consultations | On the day of enrolment.
Healthcare resource utilisation | On the day of enrolment.
Direct Healthcare costs | On the day of enrolment.

OTHER OUTCOMES:
Socioeconomic background of users | On the day of enrolment.
Subgroup analysis | From data collection with participant enrolment to the completion of panel ratings, approximately 2-3 months after participant enrolment
Condition comparison | On the day of enrolment.
Time to receiving advice | On the day of enrolment.
Time to diagnosis | From data collection with participant enrolment to the completion of the follow-up survey send out 1 week after enrolment.
Quantitative and qualitative information collected in the phone survey on demographics, health seeking behaviour and user experience with the symptom checker | Approx. 1-2 weeks after enrolment.

CONTACTS AND LOCATIONS:
Locations (1):
- Reach Digital Health (formerly Praekelt.org), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No